CLINICAL TRIAL: NCT02391636
Title: Comparison Between Carbetocin and Oxytocin in Elective Caesarean Section With High Risk of Postpartum Hemorrhage: A Randomized Controlled Trial
Brief Title: Carbetocin and Oxytocin in Elective Caesarean Section With High Risk of Postpartum Hemorrhage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ghamra Military Hospital (Other)
Collaborators: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Maged El.Sherif, Registrar of OB/GYN, Ghamra Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2015-02-17; First posted 2015-03-18 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum Hemorrhage; carbetocin; oxytocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbetocin arm (Experimental): 100 μg intravenous injection at delivery of the anterior shoulder
  Interventions: Drug: Carbetocin
- oxytocin arm (Active Comparator): 5 IU intravenous injection at delivery of the anterior shoulder
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Carbetocin — at delivery of anterior shoulder
  Other Names: Pabal
  Arms: Carbetocin arm
Drug: Oxytocin — at delivery of anterior shoulder
  Other Names: Syntocinon
  Arms: oxytocin arm

SUMMARY:
Double blinded randomized controlled study

DETAILED DESCRIPTION:
Women will be randomized into two groups using COMPUTER-GENERATED RANDOM NUMBER LIST.

264 dark colored envelops will be serially numbered containing the corresponding letter of the corresponding drug that will be used.

Group C: 132 women in the carbetocin group will receive a bolus of 100 μg intravenous injection at delivery of the anterior shoulder.

Group O: 132 women in the oxytocin group will receive 5 IU of oxytocin by slow intravenous injection at delivery of the anterior shoulder.

* All patients will receive general anaesthesia.
* Operation will be carried out by a three year registrar (at least).
* Uterus will be repaired in situ. Primary endpoint: is the amount of blood loss.
* Blood loss will be estimated using the change in Hb% and hematocrit, the actual blood loss will be calculated using the following equation:
* The actual blood loss equals the estimated blood volume X difference between the initial hematocrit and the final hematocrit / the initial hematocrit

Secondary endpoints include:

1. The need for additional uterotonic medication after carbetocin or oxytocin administration.

   - Uterine tone and Uterine fundus level (with respect to the umbilical point, UP) will be monitored during CS, at the end of CS, 2 hours, 12 hours and 24 hours after delivery

   - Additional uterotonic drugs, needed if sufficient uterine tone is not achieved within 5 minutes of oxytocin or carbetocin administration, will include: i. Ergometrine 0.5 mg by slow intravenous injection. ii. Misopristol 1000 micrograms rectally.
2. The need for blood transfusion or operative interventions related to PPH

   - The need for blood transfusion or operative intervention (B-Lynch sutures, uterine artery ligation, internal iliac artery ligation, Hysterectomy) will be considered.
3. The change in hemoglobin and hematocrit post versus pre CS

   - The drop in hemoglobin level and hematocrit will be evaluated by comparing the hemoglobin concentration on admission and 24 hours after delivery.
4. The hemodynamic adverse effects and the cost-benefit of both drugs.

ELIGIBILITY:
Inclusion Criteria:

* Multiple pregnancy
* Presence of uterine fibroid
* Previous Myomectomy
* Presence of placenta previa
* Past History of PPH
* Fetal Macrosomia
* Polyhydramnios

Exclusion Criteria:

* Hypertension
* Preeclampsia
* Cardiac, Renal, Liver diseases
* Epilepsy
* History of hypersensitivity to Carbetocin

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 264 (Actual)
Dates: Start 2015-02; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
amount of blood loss | 24 hours

SECONDARY OUTCOMES:
need for another uterotonic medication | 5 minutes
  after administration of Carbetocin or Oxytocin
need for blood transfusion or operative intervention | during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Maged M El.Sherif, Principal Investigator — Ghamra Military Hospital
Locations (1):
- Ghamra Military Hospital, Cairo, Cairo Governorate, Egypt